CLINICAL TRIAL: NCT01879176
Title: Effect of Cytokine Removal in Cardiopulmonary Bypass Patients Using the Cytosorb ™ Filter
Brief Title: Cytokine Removal in Cardiopulmonary Bypass Patients
Acronym: CytoSorb
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: CytoSorbents, Inc (Industry)
Responsible Party: Principal Investigator, Dr. Martin Bernardi, Doctor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1095/2013
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Elective Cardiac Surgical Interventions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CytoSorb (Experimental): For the intervention group, the CytoSorb filter will be installed on the CPB machine in a parallel circuit to the body circulation. The flow through the filter will be driven by a roller pump with 200ml.min-1 .
  Interventions: Device: CytoSorb
- Control (No Intervention): No filter will be installed on the CPB machine.

INTERVENTIONS:
Device: CytoSorb
  Other Names: Polymer Based Adsorption Systems; ISO 13485:2003
  Arms: CytoSorb

SUMMARY:
Cardiopulmonary bypass (CPB) surgery initiates a systemic inflammatory response induced by extrinsic (e.g. anesthesia, contact activation within the extracorporeal circuit, endotoxemia) and intrinsic (e.g. tissue damage, endothelial cell activation, ischemia-reperfusion injury of myocardium) factors. Monocytes are important players in systemic inflammation and the main producers of pro- and antiinflammatory cytokines. Monocytes activated by the extracorporeal circuit lead to a dysregulation of inflammatory homeostasis, increased levels of proinflammatory plasma mediators such as TNF-a, IL-1β, IL-6 and IL-18 are joined by antiinflammatory cytokines such as IL-10. This strong inflammatory response induces post surgical monocyte immunosuppression which is indicated by an impaired production of ex vivo LPS induced TNF-a production. Also malfunction of the peripheral circulation with increased lactate levels, pronounced fluid accumulation, increased need of vasopressors and cerebral dysfunction are observed. All of these factors may delay weaning from the ventilator, recovery of organ functions and discharge from ICU. Thus measures to decrease the inflammatory process have the potential to improve the perioperative course.

Use of cytokine adsorbing circuit during CBP has an effect on circulation cytokine levels for the first 36 hours after surgery and induces a decreased inflammatory response for up to 3 days post surgery.

DETAILED DESCRIPTION:
Patients, who have an elective cardiac surgical intervention with an expected CBP duration >120 minutes (e.g.: valve surgery, coronary artery bypass graft (CABG), combined procedures) will be enrolled to the study after given informed consent.

Patients, who decline will be asked to collect their secondary outcome data to create a "real - life" group and increase the number of patients in the control group. In this "real - life" group no additional blood samples will be taken.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgical intervention with an expected CBP duration >120 minutes

Exclusion Criteria:

* Emergency procedures
* Heart transplantation
* Elective left ventricular assist device (LVAD) implantation
* Pulmonary thromendarterectomy
* Declined informed consent
* Serum creatinine > 2mg/dl
* Body mass index < 18
* Age < 18 years
* Pregnant woman
* Receiving chemotherapy or diagnosed with any disease state (e.g., AIDS) that has produced leukopenia
* Receiving antileukocyte drugs
* Receiving TNF-α Blockers, immunosuppressive drugs (e.g. tocilizumab)
* CRP > 2mg/dl
* History of Stroke
* Bilirubin >2mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hiesmayr, MD, Study Director — Medical University of Vienna; Martin H Bernardi, MD, Principal Investigator — Medical University of Vienna; Harald Rinösl, MD, Study Chair — Medical University of Vienna; Friedrich Hoffelner, Study Chair — General Hospital of Vienna; Andreas Spittler, MD, Study Director — Medical University of Vienna; Dominik Wiedemann, MD, Study Chair — Medical University of Vienna; Philipp Opfermann, MD, Study Chair — Medical University of Vienna
Locations (1):
- Divison of Cardiothoracic Anaesthesia and Intensive Care, Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bernardi MH, Rinoesl H, Dragosits K, Ristl R, Hoffelner F, Opfermann P, Lamm C, Preissing F, Wiedemann D, Hiesmayr MJ, Spittler A. Effect of hemoadsorption during cardiopulmonary bypass surgery - a blinded, randomized, controlled pilot study using a novel adsorbent. Crit Care. 2016 Apr 9;20:96. doi: 10.1186/s13054-016-1270-0. PMID 27059056
- [Derived] Wisgrill L, Lamm C, Hell L, Thaler J, Berger A, Weiss R, Weber V, Rinoesl H, Hiesmayr MJ, Spittler A, Bernardi MH. Influence of hemoadsorption during cardiopulmonary bypass on blood vesicle count and function. J Transl Med. 2020 May 15;18(1):202. doi: 10.1186/s12967-020-02369-x. PMID 32414386

RESULTS

PARTICIPANT FLOW:
Groups:
- CytoSorb: For the intervention group, the CytoSorb filter will be installed on the CPB machine in a parallel circuit to the body circulation. The flow through the filter will be driven by a roller pump with 200ml.min-1 .
  CytoSorb
Period: Overall Study
Arm/Group | CytoSorb | Control
Started | 24 | 22
Completed | 16 | 16
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Population: Patients, who were allocated to treatment or control after randomization
Groups:
- CytoSorb: For the intervention group, the CytoSorb filter will be installed on the CPB machine in a parallel circuit to the body circulation. The flow through the filter will be driven by a roller pump with 200ml.min-1.
- Total: Total of all reporting groups
Arm/Group | CytoSorb | Control | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Full Range); unit: years] | 64 [30 to 81] | 69 [50 to 81] | 67 [30 to 81]
Gender [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  Austria | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: IL-6
Time Frame: 1. Preoperative 2. Before CBP 3. After CPB 4. 2 hours after CPB 5. 24 hours 6. 48 hours 7. 120 hours
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | CytoSorb | Control
Number analyzed (Participants) | 16 | 16
pg/ml
  Preoperative | 0 [0 to 0] | 0 [0 to 0]
  Before CPB | 0 [0 to 0] | 0 [0 to 0]
  After CPB | 62.9 [10.8 to 98.7] | 63.6 [41.2 to 154.9]
  2 hours after CPB | 120.8 [49.0 to 160.8] | 118.7 [68.4 to 255.9]
  24 hours after CPB | 111.6 [53.7 to 253.5] | 120.9 [68.0 to 198.5]
  48 hours after CPB | 89.0 [61.4 to 160.5] | 67.7 [43.7 to 134.5]
  120 hours after CPB | 0.4 [0 to 8.3] | 8.2 [0.8 to 19.4]

ADVERSE EVENTS:
Arm/Group | CytoSorb | Control
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes